CLINICAL TRIAL: NCT02705664
Title: Subject Adherence and Satisfaction for Treatment of Onychomycosis With Loceryl Nail Lacquer 5% Versus a Fungal Nail Treatment Set Containing Urea 40% Ointment and Bifonazole Cream 1%
Brief Title: Treatment of Onychomycosis With Loceryl (Amorolfine) Nail Lacquer 5% Versus a Two-course Treatment With Urea 40% Ointment and Bifonazole Cream 1%
Acronym: OPEN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RD.03.SPR.105078
Record Dates: First submitted 2016-03-07; First posted 2016-03-10 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2016-09

CONDITIONS: Foot Dermatoses
Keywords: Onychomycosis
MeSH Terms: conditions — Foot Dermatoses; Onychomycosis | interventions — Urea; bifonazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Loceryl NL (Experimental): Amorolfine hydrochloride NL 5% to be applied once weekly for 7 weeks on all affected toenails of one foot
  Interventions: Drug: Loceryl Nail Lacquer
- Urea Ointment + Bifonazole Cream (Active Comparator): On the opposite foot:
  1. Urea 40% ointment to be applied once a day under occlusion for 2-3 weeks depending on the achievement of optimal diseased toenail plates removal)
  2. Bifonazole 1% cream to be applied for 4 weeks on affected toenails (after the maximum 3-week treatment period with Urea ointment)
  Interventions: Drug: Urea Ointment; Drug: Bifonazole Cream

INTERVENTIONS:
Drug: Loceryl Nail Lacquer — Topical over entire toenail plates of affected toenails once weekly in the evening (at bed time) after having filled down affected toenails to gently remove as much as affected nails and having cleaned toenails surfaces with the provided cleansing swab
  Other Names: Loceryl NL
  Arms: Loceryl NL
Drug: Urea Ointment — Topical over the infected part of the toenails only once daily under occlusion in the evening (at bed time) after having soaked toenails in warm water and having removed the soften infected toenail plates and dried the toenails
  Other Names: Urea
  Arms: Urea Ointment + Bifonazole Cream
Drug: Bifonazole Cream — Topical, to be rubbed sparingly over the affected toenail skin (nail bed) once daily in the evening (at bed time) after having cleaned and dried thoroughly toenails
  Other Names: Bifonazole
  Arms: Urea Ointment + Bifonazole Cream

SUMMARY:
The main objective of this study is to compare subject adherence and satisfaction for two modes of treatment toenails infection (Onychomycosis) with Loceryl Nail Lacquer (Loceryl NL) and a Fungal Nail Treatment Set containing Urea 40% ointment (Urea) and Bifonazole cream 1% (Bifonazole).

DETAILED DESCRIPTION:
A total of 20 subjects are to be included in 1 site in Iceland

Methodology:

Subjects will receive following treatments on the right or left toenails:

* Loceryl Nail Lacquer (Loceryl NL) to be applied once weekly for 7 weeks on all affected toenails of one foot (including great toenail)
* Fungal Nail Treatment Set to be used on all affected toenails (including great toenail) of the opposite foot in two phases:

  * Phase I: Urea ointment (Urea) to be applied once a day under occlusion for 2-3 weeks depending on the achievement of optimal diseased toenail plates removal
  * Phase II: Bifonazole cream to (Bifonazole) be applied for 4 weeks on affected toenails (after the maximum 3-week treatment period with Urea ointment)

ELIGIBILITY:
Inclusion Criteria:

* Subjects with clinically Distal and Lateral Subungual Onychomycosis (DLSO) due to dermatophytes and/or yeast (including Candida) on at least one great toenail of each foot at screening visit,
* Subjects with less than 50% of the toenail surface area from the Distal edge with disease involvement and without matrix involvement, no dermatophytoma, streaks (spikes) or subungual hyperkeratosis > 2mm,
* Subjects should have the same number of affected toenails on both feet or no more than one additional affected toenail on one of the feet,
* Subjects with positive mycological results (direct microscopy and culture) of the most affected toenail (or great toenail) for dermatophytes or yeast (including Candida) at Baseline

Exclusion Criteria:

* Subjects with matrix involvement on the great toenails,
* Subjects with a surgical, medical condition or clinically important abnormal physical findings which might interfere with the interpretation of the objectives of the study
* Post-traumatic toenail, lichen planus, eczema, psoriasis, or other abnormalities of the nail unit, which could affect/influence the subject's compliance with the investigational products or mask the effects of treatment (cure),
* Known immunodeficiency, radiation therapy, immune suppressive drugs,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
% adherent subjects with applications | Week 7
  Percent of subjects having applied both study treatments as instructed (once a week for Loceryl NL, once a day for urea and once a day for Bifonazole)
% adherent subjects with nail preparation | Week 7
  Percent of subjects having prepared affected toenails as instructed for each product before applications:
  * For Loceryl: File down the affected toenails as required and clean toenails surface with the cleansing swab
  * For Urea: Soak toenails in warm water and remove soften infected toenails plates
  * For Bifonazole: Clean and dry thoroughly affected toenails
% Subjects satisfied to very satisfied with each study treatment at week 7 | Week 7
  Percent of subjects satisfied to very satisfied with each study treatment at week 7

CONTACTS AND LOCATIONS:
Overall Officials: Dr Sigurgeirsson, Principal Investigator — Cutis Ehf (Dermatology Center)
Locations (1):
- Principal Investigator, Reykjavik, Iceland